CLINICAL TRIAL: NCT04759053
Title: Effectiveness of Core-Needle US Guided Biopsy as Primary Tool For Diagnosis of Thyroid Nodules, A Prospective Study
Brief Title: Effectiveness of Core-Needle US Guided Biopsy as Primary Tool For Diagnosis of Thyroid Nodules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmed Aouf, Dr, Assistant lecturer of general surgery, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 124569124577
Record Dates: First submitted 2021-02-09; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Thyroid Nodule; Thyroid Diseases; Thyroid Gland; Node
Keywords: Thyroid nodule; Core needle biopsy; FNB
MeSH Terms: conditions — Thyroid Nodule; Thyroid Diseases | interventions — Biopsy, Needle

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FNB (Active Comparator)
  Interventions: Procedure: FNB; Procedure: Core biopsy
- Core biopsy (Active Comparator)
  Interventions: Procedure: FNB; Procedure: Core biopsy

INTERVENTIONS:
Procedure: FNB — Fine needle aspiration from the nodules
Procedure: Core biopsy — Core biopsy from thyroid nodules

SUMMARY:
The study aimed to determine the best intervention between Core biopsy and Fine needle aspiration in diagnosis of thyroid malignancy.

ELIGIBILITY:
Inclusion Criteria:

* patients with nodules larger than 1 cm in diameter and suspicious ultrasound criteria with TIRADS category III or higher.

Exclusion Criteria:

* Patients with a history of hemodynamic instability or inadequate coagulation profile were excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Number of samples in FNB and CNB matching the final pathology | 7 days
  Comparing number of samples in FNB and CNB that make same diagnosis as the final postoperative pathology